CLINICAL TRIAL: NCT02051790
Title: Evaluation of Reader Training Processes by Comparing Clinical Interpretations to Centralized Expert Reads
Brief Title: Evaluation of Reader Training Processes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Avid Radiopharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: 18F-AV-45-RTP01
Record Dates: First submitted 2014-01-30; First posted 2014-01-31 (Estimated); Results first posted 2015-09-28 (Estimated); Last update posted 2015-09-28 (Estimated); Status verified 2015-08

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — florbetapir

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- Clinical Practice Scans (Experimental): Approximately 250 florbetapir F 18 scans and final scan reports interpreted in a clinical setting will be collected from physicians across the country. These results will then be compared to expert panel interpretations for the same scans.
  Interventions: Drug: florbetapir F 18

INTERVENTIONS:
Drug: florbetapir F 18 — No study drug will be administered in this study - scans previously acquired in the course of clinical practice.
  Other Names: 18F-AV-45; Amyvid; florbetapir

SUMMARY:
This study is designed to evaluate the agreement between florbetapir F 18 scan interpretation in the clinic and by expert readers.

ELIGIBILITY:
Inclusion Criteria:

- Scan obtained for clinical reasons

Exclusion Criteria:

- None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 241 (Actual)
Dates: Start 2014-03; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chief Medical Officer, Study Director — Avid Radiopharmaceuticals
Locations (1):
- Research Site, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Clinical Practice Scans: 241 florbetapir F 18 scans and final scan reports interpreted in a clinical setting were collected from physicians across the country. These results were then compared to expert panel interpretations for the same scans.
  florbetapir F 18: No study drug was administered in this study - scans previously acquired in the course of clinical practice.
Period: Overall Study
Arm/Group | Clinical Practice Scans
Started | 241
Completed | 241
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Clinical Practice Scans
Number analyzed (Participants) | 241
Age, Customized [Number; unit: scans] — Age was not collected in this study.
  scans
    Age Unknown | 241
Sex/Gender, Customized [Number; unit: scans] — Gender was not collected in this study.
  scans
    Gender Unknown | 241
Region of Enrollment [Number; unit: scans] — All scans were collected from imaging centers in the US.
  scans
    United States | 241

OUTCOME MEASURES:

1. Primary Outcome: Agreement Between Expert Panel and Clinical Practice Reads
Description: Agreement between expert panel consensus scan interpretations and clinical practice reader scan interpretations was calculated as a weighted Kappa value across all cases and all clinical practice readers.
Time Frame: Scan acquired 50-60 minutes post injection
Measure: Number (95% Confidence Interval); unit: Weighted Kappa statistic
Arm/Group | Clinical Practice Scans
Number analyzed (Participants) | 241
Weighted Kappa statistic | 0.745 [0.6649 to 0.8260]

ADVERSE EVENTS:
Description: No study drug was administered in this study - scans previously acquired in the course of clinical practice, therefore no adverse event information was collected.
Arm/Group | Clinical Practice Scans
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No